CLINICAL TRIAL: NCT05379426
Title: Older Adults' Perceptions About the Impact of COVID-19 Pandemic on Their Cognitive, Emotional and Social Status: A Multicentre Mixed Methods Study in Institutions Providing Care and Supporting Services for Older Adults
Brief Title: Older Adults' Perceptions of the Impact COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Rsocialform - Geriatria, Lda (Other)
Responsible Party: Sponsor
Other Study IDs: 13052022
Record Dates: First submitted 2022-05-17; First posted 2022-05-18 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: COVID-19 Pandemic; Depression, Anxiety; Cognitive Impairment; Quality of Life; Loneliness
Keywords: older adults; COVID-19; cognitive function; executive function; mood; depression; anxiety; loneliness; quality of life
MeSH Terms: conditions — COVID-19; Depression; Anxiety Disorders; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screening tests and semi-structured interview: Battery of screening tests with semi-structured interview First, the Mini-Mental State Examination will be administered to participants to assess whether they meet the inclusion criteria and an identification code will be assigned to eligible participants. Posteriorly, a clinical psychologist will administer the Frontal Assessment Battery, Center for Epidemiologic Studies Depression Scale, Geriatric Anxiety Inventory, Loneliness Scale 3 Portuguese version, Quality of Life - Alzheimer's Disease, and will conduct a semi-structured interview about the difficulties experienced by the older adult during the pandemic period.
  Interventions: Other: Impact COVID-19 pandemic

INTERVENTIONS:
Other: Impact COVID-19 pandemic — Battery of screening tests and the semi-structured interview focusing on the difficulties experienced by the older adult during the pandemic period.

SUMMARY:
This multicentre study will be conduct in several Portuguese institutions, which provide care and supporting services for older adults, with aim to assess the impact of COVID-19 pandemic on the cognitive, emotional and social status of their beneficiaries. Initially, data on global cognitive function, executive function, mood, anxiety, loneliness, and quality of life will be collected. Secondly, a semi-structured interview will be carried out to realize and understand what were the major difficulties experienced by the older adult during the pandemic period.

DETAILED DESCRIPTION:
The pandemic COVID-19 imposed the mobilisation of institutions providing care and supporting services for older adults, and the adoption of new habits on a large scale and in a very short period of time. The need to change daily routines proved to be particularly impactful among older adults, since these citizens, due to their vulnerability to adverse health outcomes and the need for additional protection against the exposure to the risk of viral infection, were subjected to more demanding and inflexible containment measures (Organisation for Economic Co-operation and Development, 2020). The confinement measures resulted in considerable restriction of independence and access to supportive social networks, making it necessary to use compensatory solutions, such as the use of digital technologies and the resolution of emerging problems remotely. However, given that, as suggested by recent statistical data (European Commission, 2020; European Union, 2020), a large proportion of older adults do not have access to suitable equipment or lack adequate digital skills, the effective and satisfactory mobilisation of these compensatory solutions depended, in many cases, on the involvement of others. As a result, older adults saw their personal autonomy compromised and their relationships with other people highly limited. The confinement measures also resulted in the abandonment of at least some healthy living habits (moments of conviviality, cognitive stimulation activities, physical exercise and recreational activities carried out in groups, etc.), which are essential for the maintenance of physical and cognitive capacities, contributing to the increase of well-being and quality of life.

Taking into account the duration of the COVID-19 pandemic, it is necessary to understand its impact on the cognitive, emotional, and social status of older adults. Our proposal focuses on older adults who benefit from care and support services (e.g., long-term care centres, day and social centres, home support services), in which the pandemic mitigation measures were particularly rigorous, being supported by contingency plans constantly updated according to the guidelines issued by the Portuguese Directorate-General of Health and supervisory entities.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 or over.
* Native Portuguese speakers.
* Have handed in the project informed consent, duly completed and signed, after prior information.
* Communication and comprehension skills.
* Have been attending a care and support services for the older adults for at least two years.

Exclusion Criteria:

* Severe sensory and physical limitations or an acute or serious illness preventing participation in the study.
* Evidence of aggressive and disruptive behaviour, as indicated by the reference technicians of the institution where the participant attends a care and support services.
* Consumption of psychoactive substances and/or taking neuroleptics or antipsychotics in the last two months.
* Presence of a score lower than 10 points in the Mini Mental State Examination.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: In each participating institution, users who meet the inclusion criteria will be assigned to answer/fill in the assessment instruments. Prior to the enrolment in the study, informed consent will be obtained from participants after they have received information about the study. This information will include the purpose of the study, the assessment procedures adopted, the data processing procedures in accordance with current legislation, the voluntary nature of participation in the study and the right to withdraw consent at any time without affecting the services received in the institution.
Sampling Method: Non-Probability Sample
Enrollment: 880 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Cognitive functioning assessed through Mini-Mental State Examination (MMSE) | baseline
  Cognitive functioning will be assessed using the MMSE, which is a gold standard for assessing global cognitive function. Scores range from 0 to 30, with higher scores indicating better cognitive functioning.
Executive functions assessed through Frontal Assessment Battery (FAB) | baseline
  FAB assesses executive functions such as abstract thinking, mental flexibility, motor programming, interference sensibility, inhibitory control and environmental independence. Scores range between 0 - 18 points. Higher scores indicate better cognitive function.
Depressive symptomatology assessed through the Center for Epidemiologic Studies Depression Scale (CES-D) | baseline
  This instrument assesses depressive symptoms based on 20 statements classified on the frequency scale, with reference to the week prior to the assessment. Scores range between 0 and 60 points. Higher scores indicate more severe depressive symptoms.
Anxiety symptomatology assessed through the Geriatric Anxiety Inventory (GAI) | baseline
  GAI assesses, in several contexts, the severity of anxiety symptoms in older adults. It consists of 20 dichotomous response items (I agree/disagree) and refers to the subject's feelings in the week prior to the evaluation. One (1) point is assigned to each agree answer and the overall score is obtained by adding the scores of all items. Scores over 10/11 points indicate symptoms of severe anxiety.
Loneliness assessed through Loneliness Scale 3 Portuguese version (UCLA) | baseline
  UCLA is composed of 20 items. Each item is answered according to a Likert scale from 1 (never) to 4 (always). Items 1, 5, 6, 9, 10, 15, 16, 19 and 20 are inverse-scored. Scores range from 20 to 80 points. Higher scores indicate a higher level of loneliness or perceived social isolation.
Quality of life assessed through Quality of Life - Alzheimer's Disease (QoL-AD) | baseline
  The QoL-AD is used to assess quality of life. This 13-item scale assesses the quality of life in people diagnosed with dementia, gathering information from the patient about the following domains: perceived health, mood, physical condition, interpersonal relationships, hobbies, decision-making skills, and life as a whole. Scores range from 13 to 52, with higher scores indicating better quality of life.

OTHER OUTCOMES:
Sociodemographic information gathered through the sociodemographic questionnaire | baseline
  The sociodemographic questionnaire was designed specifically for this study. It gathers information about the participants' gender, age, marital status, educational level, care and support services that the participant attends, medical comorbidities, including cognitive ones, and pharmacological treatment. It will be administered to all participants.
Difficulties experienced by the older adult during the pandemic period gathered through the semi-structured interview | baseline
  The semi-structured interview was designed specifically for this study. It will gather information about the participants' difficulties experienced during the pandemic period. It will only be administered to participants with a high MMSE score, according to their educational level, and with the language ability that ensures the comprehensibility of their interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Susana I Justo Henriques, Ph.D., Principal Investigator — Health Sciences Research Unit: Nursing (UICISA: E), Nursing School of Coimbra; Elzbieta Bobrowicz Campos, Ph.D., Principal Investigator — Health Sciences Research Unit: Nursing (UICISA: E), Nursing School of Coimbra; João L Alves Apóstolo, Ph.D., Principal Investigator — Health Sciences Research Unit: Nursing (UICISA: E), Nursing School of Coimbra
Locations (58):
- Portugal (58):
  - Santa Casa da Misericórdia de Albergaria-a-Velha, Albergaria-a-Velha, Aveiro District
  - Cediara - Associação de Solidariedade Social de Ribeira de Fráguas, Albergaria-a-Velha, Aveiro District
  - Santa Casa da Misericórdia de Angra do Heroísmo, Angra do Heroísmo, Azores
  - Lar Recolhimento Jesus Maria José - Mónicas, Angra do Heroísmo, Azores
  - Santa Casa da Misericórdia da Calheta, Calheta, Azores
  - Santa Casa da Misericórdia da Horta, Horta, Azores
  - Lar D. Pedro V, Praia da Vitória, Azores
  - Centro Comunitário de São Brás, Praia da Vitória, Azores
  - Casa de Repouso João Inácio de Sousa, Velas, Azores
  - Santa Casa da Misericórdia de Vila do Porto, Vila do Porto, Azores
  - Santa Casa da Misericórdia de Mértola, Mértola, Beja District
  - ASCRA - Associação Social, Cultural e Recreativa de Apúlia, Apúlia, Braga District
  - Santa Casa da Misericórdia de Barcelos, Barcelos, Braga District
  - Centro Social da Paróquia de Vieira do Minho, Vieira do Minho, Braga District
  - Santa Casa da Misericórdia de Mirandela, Mirandela, Braganza District
  - Santa Casa da Misericórdia de Vila Velha de Rodão, Vila Velha de Rodão, Castelo Branco District
  - Santa Casa da Misericórdia da Lousã, Lousã, Coimbra District
  - Santa Casa da Misericórdia de Portimão, Portimão, Faro District
  - Associação dos Amigos de Peva, Peva, Guarda District
  - Santa Casa da Misericórdia de Alcobaça, Alcobaça, Leiria District
  - Santa Casa da Misericórdia de Alvaiázere, Alvaiázere, Leiria District
  - Santa Casa da Misericórdia de Alvorge, Alvorge, Leiria District
  - Centro Social e Paroquial Alcabideche, Alcabideche, Lisbon District
  - Associação do Hospital Civil e Misericórdia de Alhandra, Alhandra, Lisbon District
  - APOIARTE - Associação de Apoio aos Artistas, Carnide, Lisbon District
  - Centro Social Paroquial de Oeiras, Oeiras, Lisbon District
  - Associação de Socorros da Freguesia de Turcifal, Torres Vedras, Lisbon District
  - Associação de Desenvolvimento Comunitário do Funchal - Garouta do Calhau, Funchal, Madeira
  - Santa Casa da Misericórdia de Arez, Arez, Portalegre District
  - Santa Casa da Misericórdia de Avis, Avis, Portalegre District
  - Lar Júlio Alcântara Botelho, Elvas, Portalegre District
  - Lar e Centro de Dia Padre Américo, Penafiel, Porto District
  - Santa Casa da Misericórdia da Trofa, Trofa, Porto District
  - Santa Casa da Misericórdia de Rio Maior, Rio Maior, Santarém District
  - Santa Casa da Misericórdia de Caminha, Caminha, Viana do Castelo District
  - Santa Casa da Misericórdia de Ponte de Lima, Ponte de Lima, Viana do Castelo District
  - Santa Casa da Misericórdia de Vila Nova de Cerveira, Vila Nova de Cerveira, Viana do Castelo District
  - A.S.S.F.A., Abraveses, Viseu District
  - Santa Casa da Misericórdia de Tarouca, Tarouca, Viseu District
  - Santa Casa da Misericórdia de Vouzela, Vouzela, Viseu District
  - Fundação Casa do Pessoal da Segurança Social e Saúde do Distrito de Aveiro, Aveiro
  - Associação Grupo Desportivo e Social Penso Santo Estevão, Braga
  - Centro Zulmira Pereira Simões, Braga
  - Obra Social Padre Miguel, Bragança
  - Santa Casa da Misericórdia de Castelo Branco, Castelo Branco
  - Residência Sénior D. António, Castelo Branco
  - Centro Social Rocha Barros, Coimbra
  - Fundação João Bento Raimundo, Guarda
  - Centro Social Paroquial da Ilha - Obra Social da Sagrada Família, Leiria
  - Centro Social Paroquial São Mamede, Lisbon
  - Associação Casapiana de Solidariedade, Lisbon
  - Fundação AFID Diferença, Lisbon
  - Centro Comunitário e Paroquial da Ramada, Lisbon
  - Centro Social Paroquial de Oliveira do Douro, Porto
  - Associação de Solidariedade Social S. Tiago de Rebordões, Porto
  - Centro Social e Cultural de Carreço, Viana do Castelo
  - Centro Social Paroquial de Mateus, Vila Real
  - Santa Casa da Misericórdia de Montemor-o-Novo, Montemor-o-Novo, Évora District

IPD SHARING:
Plan to Share IPD: No